CLINICAL TRIAL: NCT03480230
Title: Phase II Trial of Neoadjuvant Compound 121564 Plus Platinum Doublet Chemotherapy in Non-Small Cell Lung Cancer
Brief Title: Neoadjuvant Compound 121564 Plus Platinum Doublet Chemotherapy in Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arafat Tfayli (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); Phoenix Clinical Research (Other)
Responsible Party: Sponsor-Investigator, Arafat Tfayli, Professor of Clinical Medicine, American University of Beirut Medical Center
Organization: American University of Beirut Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2017-0467; MS100070_0020 (Other Grant/Funding Number: Merck KGaA)
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Non-Small Cell Lung Cancer Stage
Keywords: Non-small cell lung cancer; Platinum doublet chemotherapy; Neoadjuvant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): 1. Non-squamous histology:
     * Compound 121564 10 mg/Kg administered over 60 minutes given intravenously every 2 weeks for 4 doses.
     * Compound 565994 500 mg/m2 administered over 10 minutes, and
     * Compound 232673 AUC=5 mg/mL/min administered over 15-60 minutes or Compound 454893 at 75 mg/m2 over 1 hour.
     * Compound 565994 and platinum are to be given on day 1 of every 3-week cycle for 3 cycles.
  2. Squamous histology:
     * Compound 121564 10 mg/Kg administered over 60 minutes every 2 weeks for 4 doses.
     * Compound 232673 AUC=5 mg/mL/min administered over 15-60 minutes or Compound 454893 at 75 mg/m2 over 1 hour on day 1 of every cycle.
     * Compound 343782 1,000 mg/m2 administered over 30 minutes on days 1 and 8 of each cycle.
     * Platinum and Compound 343782 will be given for 3 cycles.
  Interventions: Drug: Compound 121564

INTERVENTIONS:
Drug: Compound 121564 — Compound 121564 10 mg/Kg administered over 60 minutes given intravenously every 2 weeks for 4 doses plus chemotherapy depending on tumor histology.

SUMMARY:
The purpose of this study is to assess the response rate to neoadjuvant Compound 121564 plus platinum doublet chemotherapy in patients with early stage non-small cell lung cancer.

DETAILED DESCRIPTION:
Open-label, single-arm multi-center phase II trial of neoadjuvant Compound 121564 plus platinum doublet chemotherapy conducted among patients with early stage (IB, II, IIIA) non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥ 18 years.
2. Histologically confirmed NSCLC (squamous and non-squamous).
3. High-risk stage IB (tumor ≥ 4 cm in size, or grade 3, or with visceral pleura involvement), II or IIIA disease.
4. Have biopsy tissue available (fresh and archived) for PD-L1 and correlative studies testing prior to therapy.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤

1. 6) Have a life expectancy of ≥ 6 months. 7) No previous systemic anticancer therapy or surgical resection for his or her NSCLC. 8) Subject has voluntarily agreed to participate by giving written informed consent for the trial. 9) Subject must be willing and able to comply with scheduled visits, treatment schedule and laboratory testing. 10) Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to receiving the first dose of study medication. 11) Females should not be breastfeeding. 12) Female subjects of childbearing potential as well as males sexually active with women of childbearing potential must be willing to use an adequate method of contraception. 13) Have pulmonary and cardiac function testing deemed adequate for thoracic surgical intervention. 14) Have adequate organ function by meeting the following:

1. Absolute neutrophil count (ANC) ≥1,500/mcL.
2. Platelets ≥100,000/mcL.
3. Hemoglobin ≥9 g/dL.
4. Serum creatinine ≤1.5 X upper limit of normal (ULN) OR calculated creatinine clearance (CrCl) (GFR can also be used in place of creatinine or CrCl) ≥60 mL/min for subjects with creatinine levels > 1.5 X institutional ULN.
5. Serum total bilirubin ≤ ULN.
6. AST (SGOT) and ALT (SGPT) ≤ 1.5 X ULN.
7. Alkaline phosphatase ≤ 2.5 X ULN.
8. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless the subject is receiving anticoagulant therapy.
9. Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless the subject is receiving anticoagulant therapy.

Exclusion Criteria:

1. Subject deemed unfit for surgery (by pulmonary or cardiac assessment).
2. Subject with known autoimmune disease that has required systemic therapy in the last 2 years.
3. Prior organ transplantation including allogenic stem-cell transplantation.
4. Clinically significant (i.e. active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
5. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
6. Subject on immunosuppressive therapy or corticosteroids within 14 days prior to starting study drugs.
7. Subject with interstitial lung disease that is symptomatic or history of pneumonitis that required oral or systemic glucocorticoids to manage.
8. Subject must have recovered from the effects of major surgery or significant trauma at least 14 days prior to therapy.
9. Subject with previous malignancies are excluded unless complete remission was achieved at least 2 years prior to therapy.
10. Other active malignancy requiring concurrent intervention.
11. Subject with active infection requiring systemic therapy.
12. Subject with known history of testing positive for human immunodeficiency virus (HIV) or known to have acquired immunodeficiency syndrome (AIDS).
13. Subject has known active hepatitis B or C.
14. Vaccination within 4 weeks of the first dose of Compound 121564 and while on trials is prohibited except for administration of inactivated vaccines.
15. Subject is pregnant or breastfeeding.
16. Subject has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Subject previously had a severe hypersensitivity reaction to any of the study drugs.
18. Subject is currently participating and receiving study therapy from another clinical trial.
19. Subject had prior treatment with any other anti-PD-1, or PD-L1 or PD-L2 agent or an antibody targeting other immuno-regulatory receptors or mechanisms.
20. Patient who is not willing to sign the consent form.
21. Legal incapacity or limited legal capacity patients receiving other oncology specific medication not authorized in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-26 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) as assessed by RECIST 1.1 criteria | At week 9
  To assess the overall response rate (ORR) of patients receiving neoadjuvant Compound 121564 plus platinum doublet chemotherapy based on RECIST 1.1 criteria

SECONDARY OUTCOMES:
Pathologic complete response rate | At 12 weeks
  To assess the pathologic complete response rate in patients receiving combination Compound 121564 and chemotherapy.
Major pathologic response rate (<10% viable tumor cells) | At 12 weeks
  To assess the major pathologic response rate (<10% viable tumor cells) in patients receiving combination Compound 121564 and chemotherapy.
Progression-Free Survival (PFS) | At 1, 2 and 3 years
  To assess progression-free survival (PFS) at 1, 2 and 3 years in patients receiving a combination of Compound 121564 plus platinum doublet chemotherapy.
Overall Survival (OS) | At 1, 2 and 3 years
  To assess overall survival (OS) in patients receiving a combination of Compound 121564 plus platinum doublet chemotherapy.
Overall Response Rate (ORR) as assessed by RECIST 1.1 criteria in enrolled squamous vs. non-squamous lung cancer patients | At week 9
  To compare the ORR in enrolled squamous vs. non-squamous lung cancer patients receiving the proposed treatment regimen.
Progression-Free Survival (PFS) in enrolled squamous vs. non-squamous lung cancer patients | At 1, 2 and 3 years
  To compare the PFS in enrolled squamous vs. non-squamous lung cancer patients receiving the proposed treatment regimen.
Overall Survival (OS) in enrolled squamous vs. non-squamous lung cancer patients | At 1, 2 and 3 years
  To compare the OS in enrolled squamous vs. non-squamous lung cancer patients receiving the proposed treatment regimen.
Patient-related outcomes Quality of Life assessment using the questionnaire for functional assessment of cancer therapy for patients with lung cancer (FACT-L version 4) | At week 9
  To assess patient-related outcomes in patients receiving a combination of Compound 121564 plus platinum doublet chemotherapy.
Number of participants with treatment-related adverse events as assessed by CTCAE v 4.0 | With every administration
  To assess the tolerability of the proposed treatment regimen in the cohort of patient enrolled.
Overall Response Rate (ORR) as assessed by RECIST 1.1 criteria in patients with 50% or more PD-L1 vs. patients with less than 50% PD-L1 | At week 9
  To analyze as exploratory analysis the ORR in patients with 50% or more PD-L1 expression level vs. patients with less than 50% PD-L1 expression level receiving the proposed treatment regimen.
Progression-Free Survival (PFS) in patients with 50% or more PD-L1 vs. patients with less than 50% PD-L1 | At 1, 2 and 3 years
  To analyze as exploratory analysis the PFS in patients with 50% or more PD-L1 expression level vs. patients with less than 50% PD-L1 expression level receiving the proposed treatment regimen.
Overall Survival (OS) in patients with 50% or more PD-L1 vs. patients with less than 50% PD-L1 | At 1, 2 and 3 years
  To analyze as exploratory analysis the OS in patients with 50% or more PD-L1 expression level vs. patients with less than 50% PD-L1 expression level receiving the proposed treatment regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Arafat H Tfayli, MD, Principal Investigator — American University of Beirut Medical Center
Locations (5):
- King Hussein Cancer Center, Amman, Jordan
- Lebanon (4):
  - American University of Beirut Medical Center, Beirut
  - Bellevue Medical Center, Beirut
  - Lebanese American University Medical Center-Rizk Hospital, Beirut
  - Hammoud Hospital University Medical Center, Sidon

IPD SHARING:
Plan to Share IPD: Undecided